CLINICAL TRIAL: NCT00809042
Title: The Effect of Combination Therapy of Hydroxyurea With L- Carnitine and Magnesium Chloride on he-Matologic Parameters and Cardiac Function of β-Thalassemia Intermedia Patients.
Brief Title: Combination Therapy of Hydroxyurea With L-Carnitine and Magnesium Chloride in Thalassemia Intermedia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Mehran Karimi, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: SHaghpanah; 3342
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: β-Thalassemia Intermedia
Keywords: Hydroxyurea; magnesium chloride; L-carnitine; β-thalassemia intermedia
MeSH Terms: interventions — Hydroxyurea; Carnitine; Magnesium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Hydroxyurea
  Interventions: Drug: hydroxyurea
- 2 (Active Comparator): L-carnitine and hydroxyurea
  Interventions: Drug: L-carnitine and hydroxyurea
- 4 (Active Comparator): L-carnitine , magnesium chloride and hydroxyurea
  Interventions: Drug: hydroxyurea,L-carnitine and magnesium chloride
- 3 (Active Comparator): magnesium chloride and hydroxyurea
  Interventions: Drug: hydroxyurea and magnesium chloride

INTERVENTIONS:
Drug: hydroxyurea — Hydroxyurea (500 mg capsules) was administered in a single dose at a mean of 10/mg/kg/day (range8-12mg/kg/day).
  Arms: 1
Drug: L-carnitine and hydroxyurea — Hydroxyurea (500 mg capsules) was administered in a single dose at a mean of 10/mg/kg/day (range8-12mg/kg/day). L-carnitine (Minoo, Iran, 250 mg tablets) was administered in divided doses (50mg/kg/day).
  Arms: 2
Drug: hydroxyurea and magnesium chloride — Hydroxyurea (500 mg capsules) was administered in a single dose at a mean of 10/mg/kg/day (range8-12mg/kg/day). Magnesium chloride powder ( tabib tajhiz nik, Iran) was formulated into suspension; each ml containing 1meq magnesium chloride. It was administered in divided doses at 0.6meq/kg/day.
  Arms: 3
Drug: hydroxyurea,L-carnitine and magnesium chloride — Hydroxyurea (500 mg capsules) was administered in a single dose at a mean of 10/mg/kg/day (range8-12mg/kg/day). L-carnitine (Minoo, Iran, 250 mg tablets) was administered in divided doses (50mg/kg/day). Magnesium chloride powder ( tabib tajhiz nik, Iran) was formulated into suspension; each ml containing 1meq magnesium chloride. It was administered in divided doses at 0.6meq/kg/day
  Arms: 4

SUMMARY:
The purpose of this study is determination of the efficacy of combination of hydroxyurea with L-carnitine or magnesium in improving hematologic parameters and cardiac status in patients with β-thalassemia intermedia in comparison with hydroxyurea alone .

ELIGIBILITY:
Inclusion Criteria:

* Beta thalassemia intermedia patients with mean hemoglobin level >= 7gr/dl, need to blood transfusion with more than 6 months interval or no need to blood transfusion

Exclusion Criteria:

* Hypothyroidism
* Hypoparathyroidism
* Diabetes mellitus
* Hepatitis B and C
* Positive tests for human immunodeficiency virus
* Any cardiac symptoms or receiving drug for cardiac disease
* Presence of other hemoglobinopathies except thalassemia intermedia and pregnant or lactating womens

Ages: 4 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Hematologic Parameters | monthly

SECONDARY OUTCOMES:
echocardiographic parameters | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Karimi, Full Professor, Principal Investigator — Hematology Research Center of Shiraz University of Medical Sciences
Locations (1):
- Hematology Research Center of Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Foong WC, Loh CK, Ho JJ, Lau DS. Foetal haemoglobin inducers for reducing blood transfusion in non-transfusion-dependent beta-thalassaemias. Cochrane Database Syst Rev. 2023 Jan 13;1(1):CD013767. doi: 10.1002/14651858.CD013767.pub2. PMID 36637054